CLINICAL TRIAL: NCT01315418
Title: Effect of the Consumption of a Fermented Milk on Common Infections in Adults Submitted to Multi-stressor Situation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU201
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Last update posted 2016-11-25 (Estimated); Status verified 2016-11

CONDITIONS: Upper Respiratory Tract Infections; Rhinopharyngitis; Sore Throat; Sinusitis; Otitis; Lower Respiratory Tract Infections; Bronchitis; Pneumopathy; Flu; Flu-like Syndromes; Gastroenteritis
Keywords: Probiotic - Lactobacillus casei DN-114 001 - dairy product -; infections - firemen; Common infectious diseases, occuring in healthy subjects,; including upper respiratory tract infections (defined as; rhinopharyngitis, sore throat, sinusitis and otitis); lower respiratory tract infections (defined as bronchitis; pneumopathy and flu and flu-like syndromes); gastrointestinal tract infection defined as gastroenteritis
MeSH Terms: conditions — Respiratory Tract Infections; Nasopharyngitis; Pharyngitis; Sinusitis; Otitis; Bronchitis; Lung Diseases; Influenza, Human; Gastroenteritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Active Comparator)
  Interventions: Other: 1-Fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel®)
- 2 = Control product (Sham Comparator)
  Interventions: Other: 2-Non fermented dairy product (control)

INTERVENTIONS:
Other: 1-Fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel®)
  Arms: 1 = Tested product
Other: 2-Non fermented dairy product (control)
  Arms: 2 = Control product

SUMMARY:
This multicentric, randomized, double-blind and controlled study aims to examine the effect of a fermented dairy product containing the probiotic Lactobacillus casei DN-114 001 (Actimel® = tested product) on the incidence of respiratory and gastro-intestinal common infectious diseases (cumulated number of infections during the intervention period: primary criteria), and on the Quality of Life in adults submitted to multi-stressor situation. Volunteers received either 200g/day of tested product (N=121) or control product (N=118) for 7-weeks.

ELIGIBILITY:
Inclusion Criteria:

* male and female aged 18-29 years
* attending 7 weeks of firemen training school
* a 19 to 29 kg/m2 body mass index
* found medically healthy (in particular, free of respiratory and GI tract symptoms)
* agreeing to a written informed consent, and who appreciates dairy products and multi-fruit flavour.

Exclusion Criteria:

* Subject who is not reading and writing French, or not understanding informed consent or study protocol
* subject with allergy or hypersensitivity to milk proteins or dairy foods components (ex: lactose), or with any known food or respiratory allergy;
* subject presenting a severe evolutive or chronic pathology (Ex: cancer, tuberculosis, Crohn disease, cirrhosis, multiple sclerosis, Type I diabetes…) or any past or actual health condition that may interfere with the outcome of the study (Ex: HIV, Chemotherapy, malabsorption, ulcer, celiac disease…)
* subject having experienced any infectious disease during the last 7 days
* subject with current diarrhoea or constipation
* subject who is frequently using laxatives or who has been using laxatives during the week prior his participation to the study
* subject who was under artificial nutrition, had gastro-intestinal surgery or any intervention requiring general anaesthesia the last 2 months prior to his participation to the study
* subject with special medicated diet (obesity, anorexia, metabolic pathology, nutritional complementation…) or with eating disorders (anorexia, bulimia, alcoholism…)
* subject currently receiving, or who has received during the last months, systemic treatment or topical treatment likely to interfere with evaluation of the study parameters: antibiotics, antiseptics,antifungal, corticoids, vaccines, anti-histaminic molecules, non-corticoid anti-inflammatory substances, immunosuppressant treatment…
* subject already enrolled in another clinical study, or currently under an exemption period from a previous study
* female subject who is currently pregnant or breast-feeding, or willing to become pregnant during the 2 coming months after enrolment in the study
* subject in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 239 (Actual)
Dates: Start 2006-12; Primary Completion 2007-05 (Actual); Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Médecin-chef du Groupement Formation Instruction, Villeneuve-Saint-Georges, France